CLINICAL TRIAL: NCT06586255
Title: Phase I Safety Trial of Concurrent Adjuvant Immunotherapy and Radiation Therapy for the Treatment of Urothelial Bladder Cancer
Brief Title: Adjuvant Concurrent Immunotherapy and Radiotherapy for the Treatment of Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 16824; 856691 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma Bladder; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Concurrent Immunotherapy and Radiation Therapy (Experimental): Subjects will receive the standard of care procedures and follow-up for immunotherapy and radiation therapy. The part of this study that is research is receiving both of these treatments at the same time.
  Interventions: Radiation: Concurrent Immunotherapy and Radiation Therapy

INTERVENTIONS:
Radiation: Concurrent Immunotherapy and Radiation Therapy — Radiation therapy will begin between 12 to 18 weeks from the start of adjuvant nivolumab. Patients will receive radiation therapy for about 6 weeks.

SUMMARY:
The primary objective of this Phase I study is to establish the safety of adjuvant concurrent immunotherapy and radiation therapy for urothelial bladder cancer.

DETAILED DESCRIPTION:
Patients in this study will receive the standard of care procedures and follow-up for immunotherapy and radiation therapy. The part of this study that is research is receiving both of these treatments at the same time. Safety will be based on acute toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pure or mixed variant urothelial carcinoma

  o Allowable mixed variant subtypes include:
  * squamous differentiation
  * glandular differentiation
  * nested pattern
  * microcystic
  * micropapillary
  * lymphoepthelioma-like
  * plasmacytoid and lymphoma-like
  * sarcomatoid/carcinosarcoma
  * giant cell
  * trophoblastic differentiation
  * clear cell
  * lipid cell
  * undifferentiated
* Radical cystectomy and pelvic lymph node dissection within the prior 48 weeks
* Pathologic T3 or higher stage disease, any N, M0 (AJCC, 7th Ed., Appendix C)
* Receiving adjuvant checkpoint inhibitor therapy
* No clinical evidence of residual or recurrent disease based on the following minimum diagnostic work-up within 3 months of a patient's consent to participate.

  * History and physical examination
  * Chest imaging by x-ray (PA and lateral views), CT scan (with or without IV contrast) or as part of a FDG PET-CT;
  * Axial abdominal and pelvic imaging by MRI (preferably with gadolinium), CT scan (with or without IV contrast) or as part of a FDG PET-CT;
  * Patients with microscopically involved (positive) surgical margins, but no grossly evident residual disease by imaging or physical exam are eligible.
* The patient is a candidate for definitive external beam radiotherapy;

  * No prior radiotherapy to the region of study;
  * No inflammatory bowel disease, active collagen vascular or connective tissue disorders, and no other medical or social contraindications to radiotherapy, as determined by a participating radiation oncologist;
* Age greater than or equal to 18 years
* ECOG performance status: 0-2
* Concurrent non-investigational medications will be permitted
* In addition to diagnostic staging scan, patient will be considered eligible only if he/she has a CT simulation scan that does not show any evidence of recurrent disease
* Informed consent: Patients must have the ability to understand and be willing to sign the study-specific informed consent indicating their understanding of the investigational nature and the risks of this study before any of the protocol related studies are performed (this does not include routine laboratory testing or imaging studies required to establish study eligibility)

Exclusion Criteria:

* Urinary diversion with an orthotopic neobladder
* History of inflammatory bowel disease
* Prior partial or complete small bowel obstruction either before or after radical cystectomy
* Prior radiotherapy to the pelvis;

  o Prior radiation therapy for a different cancer or disease process is allowed, provided there will be no overlap of radiation therapy fields between the participant's prior and current course of radiation therapy, radiotherapy was completed more than four weeks from enrolling in this study.
* Planned concurrent chemotherapy or other investigational drug to be given with radiation treatments

  o Prior chemotherapy or investigational drug for bladder cancer or a different cancer is allowed, provided that:
  * The therapy was completed more than two weeks prior to the start of adjuvant pelvic radiation
  * The participant has recovered to Grade ≤1 toxicity from agents previously administered, excluding toxicities that would not be expected to impact eligibility for radiation therapy including but not limited to neuropathy, alopecia and hearing loss.
* Subtotal surgical resection with clinically evident residual disease by physical exam or axial imaging.
* Prior or concurrent second invasive malignancy that, in the judgment of the investigator, may affect interpretation of the results.
* Known severe, active co-morbidity, defined as follows:

  o Any clinically significant unrelated systemic illness, medical condition, or other factor, which at the discretion of the Principal Investigators, would interfere in the safe and timely completion of study procedures, compromise the patient's ability to tolerate the protocol therapy, or is likely to interfere with the study procedures or results.
* Patients who experienced Grade 3+ GI toxicity due to surgery or nivolumab prior to enrollment in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety of concurrent adjuvant immunotherapy and radiation therapy | Within 18 weeks from start of radiation therapy
  The primary study endpoint is acute grade 3 or higher pelvic radiation related toxicity. A toxicity will be classified as related to pelvic radiation if the toxicity involves or is the result of effects on tissues that are within the 50% isodose bath of the radiation treatment as defined on the radiation treatment planning simulation scan. Toxicities will be graded by CTCAE Version 5.0.
  Concurrent adjuvant immunotherapy and radiation will be deemed safe if it is likely (i.e. a posterior probability of 50% or greater) that the acute grade 3 or higher pelvic radiation related toxicity rate is <20%.

CONTACTS AND LOCATIONS:
Overall Officials: John Christodouleas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No